CLINICAL TRIAL: NCT02491515
Title: Effects of Denosumab Therapy for Japanese Osteoporotic Patients
Brief Title: Effects of Denosumab Therapy for Japanese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomidahama Hospital (Other)
Responsible Party: Principal Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Other Study IDs: IRB9-2
Record Dates: First submitted 2015-06-27; First posted 2015-07-08 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; BMD; denosumab; previous therapy
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Denosumab — every 6 month injection
  Other Names: Prolia

SUMMARY:
In this study, the investigators would like to analyze the bone mineral density (BMD) , bone turnover makers, and fracture prevention effects of denosumab in Japanese patients under clinical practice. The participants are treated in the investigators hospital, who are under severe osteoporotic condition.

The main objective of this study is to investigate effects of denosumab. The researchers also investigate the effects of Effects of previous osteoporotic therapy to denosumab treatment. In this study, the investigators analyse the determinants of subsequent BMD increase and fracture preventing effect by teriparatide.

DETAILED DESCRIPTION:
Registry criteria: Patients treated in the investigators hospital using denosumab. Enrolled patients are severe osteoporosis; more than two previous osteoporotic fractures, low BMD (< young adult mean 65%).

Interventions: blood analyses and dual-energy X-ray absorptiometry (DXA) every 4 months Informed consent: Written informed consent will be obtained. Sample size: Five-hundreds participants

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients

Exclusion Criteria:

* cancer, hypercalcemia, etc (i.e. patients who could not use denosumab)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporotic patients who admit to our hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
BMD increase by denosumab in Japanese | Up to 48 months
  The investigators evaluate BMD increase by denosmab in Japanese patients.

SECONDARY OUTCOMES:
The determinants related to BMD increase and fracture prevention for denosumab treatment | Up to 48 months
  The investigators evaluated lumbar and femoral neck BMD. The investigators evaluated baseline patients characteristics. The investigators will evaluate the relationship between BMD increase or fracture and patients characteristics using univariate and multivariate analysis.
Effects of previous therapy to denosumab | Up to 48 months
  The investigators evaluate effects of previous osteoporosis treatment to denosumab in BMD increase and bone turnover marker response using univariate and multivariate analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Niimi, MD, Study Director — Tomidahama Hospital
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan